CLINICAL TRIAL: NCT04411927
Title: Impact of Chronic Kidney Disease on Postural Stability in Children: A Cross-sectional Observational Study
Brief Title: Impact of Chronic Kidney Disease on Postural Stability in Children
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Mahmoud Abd-elmonem, Amira Abd-elmonem, assist Prof. Physiacl therapy for pediatric department, faculty of physical therapy , Cairo university, Cairo University
Other Study IDs: children with CKD
Record Dates: First submitted 2020-05-18; First posted 2020-06-02 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Chronic Kidney Diseases
Keywords: Balance; Chronic kidney disease; HUMAC balance system; Postural stability
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- control group: this group included 25 typically developed children
  Interventions: Other: assessment of postural stability
- on-heamodialysis group: this group included children with CKD on-heamodialysis treatment
  Interventions: Other: assessment of postural stability
- non-dialysis group: this group included children with CKD who don't require dialysis
  Interventions: Other: assessment of postural stability

INTERVENTIONS:
Other: assessment of postural stability — assessment of postural stability

SUMMARY:
Background: Chronic kidney disease is associated with comorbid conditions that result in physical impairments.

Objectives: Investigate the impact of chronic kidney disease (CKD) on postural stability in children compared with age matched typically developing children using Human Assessment Computer (HUMAC) balance system.

Design: An observational design (cross-sectional study). Settings: The assessment procedures were conducted at the Nephrology Unit, Zagazig University Hospitals.

Participants: Seventy-five children, age ranged from 8 to 15 years represented three groups of equal numbers; control group (typically developed), non-dialysis (stage 3 and 4) and hemodialysis group.

Outcome measures: The HUMAC balance system was used to assess the limits of stability, center of pressure and sensory organization and balance.

DETAILED DESCRIPTION:
Methods Study design This study is an observational cross-sectional design (prospective database study).

Participants and setting Participants included children with CKD extracted from a data set of 731 individuals with CKD diagnoses, who receive regular medical follow-up/hemodialysis at Nephrology Unit, Zagazig University Hospitals. The study was conducted from January 2018 to January 2020 in accordance with the Declaration of Helsinki (Code of Ethics of the World Medical Association). The study protocol was approved by the Ethical committee of the Faculty of Physical Therapy, Cairo University, Egypt (No.P.T.REC/012/002169). Children's par-ticipation was authorized by a signed written consent form with parent's/legal guardian's acceptance for participation before starting the study procedures.

Participants Fifty eligible volunteer children with CKD were recruited from Nephrology Unit, Zagazig University Hospitals to be enrolled in this study and allocated into either hemodialysis (on hemodialysis) or non-dialysis group (children at stage 3 and 4).

Eligible criteria:

* Medically diagnosed with CKD (regardless of medical history),
* Age ranged from eight to fifteen years,
* Both genders

Participants were excluded if they had:

* Communication problems such as intellectual disability, autism, Down syndrome, or cerebral palsy,
* Significant visual or hearing problems,
* Any neurological and/or musculoskeletal disorders which influence postural stability,
* Chronic cardiovascular or pulmonary disorders. Twenty-five volunteer typically developed age matched group were enrolled as control group.

Basic demographic and clinical information Demographics and physical characteristics (age, sex, weight, height) and clinical data (renal function test, recent hematology and blood chemistry counts, co-morbidity, and medication) were recorded from medical reports to confirm diagnosis.

Study power and sample size Sample size was predestined before conducting the study by G*POWER statistical software (Franz Faul, Universitat Kiel, Germany; version 3.1.9.2) [F tests- ANOVA: Fixed effects, one-way, α=0.05, β=0.2, and large effect size] with the number of groups=3, giving a total number of 66 participants to be recruited in this study.

2.5. Outcome measures The Human Assessment Computer (HUMAC) Balance System, primarily being part of a video game appliance (Wii Balance Board), is a distinct technology used in assessment and rehabilitation of postural control. It is an affordable, portable and prevalent obtainable force plate provides the patient and tester with visual feedback as well as numerical data. The system displays several reporting options with objective datum providing clinicians with comprehensive case progression which is used for baseline and follow-up analysis with eight programs to choose from (HUMAC balance, 2017; Blosch et al., 2019). The HUMAC-type technology has been found to detect more imbalances than traditional tests (Merchant-Borna et al., 2017). In the current study limits of stability, COP and the Clinical Test of Sensory Organization and Balance (CTSIB) were assessed. Each child in the three study groups performed three trials and the mean value was estimated for each test.

2.5.1. Limits of Stability test: Limits of stability are known as the furthest distance a subject is capable to shift his/her COP in different directions whilst keeping the configuration of the BOS and adjust the body position. This commonly requires the use of a force plate that records COP movement and a visual feedback that serves to maximize COP displacement in certain directions (Lemay et al., 2014). During this test, the participant is instructed to shift the round cursor on the screen (the COP) to the highlighted target. As he/she remains in the target for the hold time, this target point is deactivated and should move between the center targets to each surrounding target in a random order. A count-up timer displays the total test time. He/she must return to the center target after each outer target. The test was conducted at two levels 4 and 6. At level 4; this is considered as simple test compared with level 6; the distance between center targets to each surrounding target is relatively small. On the other hand, at level 6 the distance between center targets to each surrounding target is larger.

2.5.2. Center of pressure test This test is used to measure the variation in a subject's COP and displays his/her Right/Left and Anterior/Posterior weight distribution. In the current study, the COP test variables recorded were the stability score and path length.

* Stability test: It measures the participant's ability to stabilize his/her balance at locations around their neutral position. Results are reported as the percent of time a subject holds his COP in each of the eight flashing targets in clockwise order (right/left and anterior/posterior weight distribution). These targets are eight specific points in which the current target flashes green when the participant is on-target and flashes yellow when he is off-target. The HUMAC system provides a counts-down of the hold time to inform the participant when he/she should move to the next target. In addition, the system provides variety of levels based on the distance from the center to the farthest target.
* Path length: The COP path length represents the COP displacement in which lower values indicate better performance (Ju-Hyeong et al., 2020).

2.5.3. Clinical Test of Sensory Organization and Balance: It is sometimes referred as the Romberg or Foam and Dome test. It is used to test how a participant's vestibular, somatosensory and visual systems integrate in the conditions of open and closed eyes compared to a normal population. The CTSIB protocol typically uses four conditions including eyes closed soft surface (ECSS); eyes closed firm surface (ECFS); eyes open soft surface (EOSS); Eye open soft surface (EOSS) and eyes open firm surface (EOFS). The participant was instructed to stand in a neutral position with the arms at body sides. Each participant went through a series of the four tests, which were each 30 seconds long. As participants completed the test, the board monitored their COG to determine their stability and path length. The requirements of the assessment were clearly demonstrated to all children. The assessment procedures were administered following the HUMAC Balance System manual detailed instructions. All participants performed three trials of each test, each lasting 30 seconds to determine the stability score and path length.

ELIGIBILITY:
Inclusion Criteria:

* Medically diagnosed with CKD (regardless of medical history),
* Age ranged from eight to fifteen years,
* Both genders

Exclusion Criteria:

Participants were excluded if they had:

* Communication problems such as intellectual disability, autism, Down syndrome, or cerebral palsy,
* Significant visual or hearing problems,
* Any neurological and/or musculoskeletal disorders which influence postural stability,
* Chronic cardiovascular or pulmonary disorders.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Fifty eligible volunteer children with CKD were recruited from Nephrology Unit, Zagazig University Hospitals to be enrolled in this study and allocated into either hemodialysis (on hemodialysis) or non-dialysis group (children at stage 3 and 4).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
limits of stability test | from January 2018 to January 2020
  it was measured by the HUMAC. higher scores indicate good balance
center of pressure (COP) test | from January 2018 to January 2020
  It was measured by the HUMAC balance system. COP is represented by
  1. path length higher scores indicate poor balance
  2. stability score with higher results indicate good balance
Clinical Test of Sensory Organization and Balance | from January 2018 to January 2020
  it was measured by the HUMAc balance system to represent the ability of the child to keep balance while standing on firm and solid surfaces alternatively with eyes open and then eyes closed

CONTACTS AND LOCATIONS:
Overall Officials: Nanees E Mohamed, Study Chair — Cairo University; Faika S Arab, Study Director — zagazieg university, Egypt; Nourhan M Baiomy, Principal Investigator — Cairo university, Egypt
Locations (1):
- faculty of physical therapy, Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided